CLINICAL TRIAL: NCT06956989
Title: Lower Urinary Tract Symptoms in Transmasculine Patients Undergoing Metoidioplasty and Their Acceptability of Pelvic Floor Muscle Training Assessed by a Pelvic, Obstetric and Gynaecological Physiotherapist
Acronym: LUTS-POGP
Status: Not yet recruiting | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 336081
Record Dates: First submitted 2025-04-07; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Lower Urinary Tract Symptoms; Transgenderism
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Lower urinary tract symptoms in transmasculine patients undergoing metoidioplasty and their acceptability of pelvic floor muscle training assessed by a Pelvic, Obstetric and Gynaecological Physiotherapist.

Study Design

Prospective observational pilot study

Study Participants

Transmasculine patients undergoing metoidioplasty

Planned Sample Size

50

Planned Study Period

2025/26

Objectives

Understand the acceptability of first-line pelvic floor muscle training (PFMT) treatment in transmasculine patients undergoing metoidioplasty

Background incidence of lower urinary tract symptoms (LUTS) in transmasculine patients undergoing surgery

Endpoints

Acceptability of PFMT questionnaire

International Prostate Symptom Score (I-PSS) and International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF) questionnaires and uroflowmetry

ELIGIBILITY:
Inclusion Criteria:

Have capacity to consent.

Diagnosis of gender dysphoria and have lived in a gender role that is congruent to their gender identity for minimum of 12 months.

Transmasculine patients referred to CCGS for masculinising lower genital reconstructive surgery having received two signatures confirming suitability for reconstructive surgery.

Undergoing metoidioplasty/phalloplasty.

Age >17 years old.

On systemic testosterone therapy for more than 12 months.

Exclusion Criteria:

* Age less than 18 years.

Not undergoing metoidioplasty/phalloplasty.

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Transgender men
Study Population: Study participants will be transmasculine patients undergoing metoidioplasty
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Understand the acceptability of first-line PFMT treatment in transmasculine patients undergoing metoidioplasty | Baseline, 6 weeks, 12 weeks, 6 months post operatively
  Acceptability of pelvic floor muscle training questionnaire - bespoke unvalidated qualitative questionnaire looking at acceptability of different PFMT techniques on a 0-10 VAS scale. Zero not acceptable, ten very acceptable.
  International prostate symptom score. Seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form questionnaires. Question items: Frequency or urinary incontinence, Amount of leakage, Overall impact of urinary incontinence, Self-diagnostic item. Scoring scale: 0-21. Higher score = worse symptoms.
  Uroflowmetry - baseline QMAX vs QMAX post procedure.
Background incidence of LUTS in transmasculine patients undergoing surgery | Baseline, 6 weeks, 12 weeks, 6 months post operatively
  Acceptability of pelvic floor muscle training questionnaire - bespoke unvalidated qualitative questionnaire looking at acceptability of different PFMT techniques on a 0-10 VAS scale. Zero not acceptable, ten very acceptable.
  International prostate symptom score. Seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form questionnaires. Question items: Frequency or urinary incontinence, Amount of leakage, Overall impact of urinary incontinence, Self-diagnostic item. Scoring scale: 0-21. Higher score = worse symptoms.
  Uroflowmetry - baseline QMAX vs QMAX post procedure.

SECONDARY OUTCOMES:
How well do the I-PSS and ICIQ SF function as measures of LUTS and LUTS specific Quality of Life (QoL) for transmen? | Baseline, 6 weeks, 12 weeks, 6 months post operatively
  Acceptability of pelvic floor muscle training questionnaire - bespoke unvalidated qualitative questionnaire looking at acceptability of different PFMT techniques on a 0-10 VAS scale. Zero not acceptable, ten very acceptable.
  International prostate symptom score. Seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form questionnaires. Question items: Frequency or urinary incontinence, Amount of leakage, Overall impact of urinary incontinence, Self-diagnostic item. Scoring scale: 0-21. Higher score = worse symptoms.
  Uroflowmetry - baseline QMAX vs QMAX post procedure.
How do subjective LUTS / objective voiding dysfunction (VD) change after metoidioplasty / vaginectomy / urethral hook up? | Baseline, 6 weeks, 12 weeks, 6 months post operatively
  Acceptability of pelvic floor muscle training questionnaire - bespoke unvalidated qualitative questionnaire looking at acceptability of different PFMT techniques on a 0-10 VAS scale. Zero not acceptable, ten very acceptable.
  International prostate symptom score. Seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form questionnaires. Question items: Frequency or urinary incontinence, Amount of leakage, Overall impact of urinary incontinence, Self-diagnostic item. Scoring scale: 0-21. Higher score = worse symptoms.
  Uroflowmetry - baseline QMAX vs QMAX post procedure.

IPD SHARING:
Plan to Share IPD: Undecided